CLINICAL TRIAL: NCT02193919
Title: A Single-Center, Prospective, Single-Blind, Pilot Study to Compare the Effect of Diet in Overweight or Obese Patients With Psoriasis on Light Therapy
Brief Title: A Single-Center, Prospective, Pilot Study to Compare the Effect of Diet in Overweight or Obese Patients With Psoriasis on Light Therapy
Status: Completed | Type: Observational
Sponsor: Bagel, Jerry, M.D. (Individual)
Responsible Party: Principal Investigator, Jerry Bagel MD, Director, Bagel, Jerry, M.D.
Other Study IDs: PO-001
Record Dates: First submitted 2013-02-04; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- cohort 1 placebo + UVB: cohort 1 placebo + UVB
- South Beach Diet + UVB: South Beach DIet + UVB
- Ornish Diet + UVB: Ornish Diet + UVB

SUMMARY:
Weight loss may help psoriasis. Phototherapy helps psoriasis. Combining the two treatments may help even more. Determining if a high protein diet vs a low protein diet results in improving psoriais may help lead to future dietary effects on psoriasis therapy

ELIGIBILITY:
Inclusion Criteria:

* PSA greater 10
* BMI greater than 30

Exclusion Criteria:

* PSA less than 10
* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients, males, females, over 18 yo with moderate-to-severe psoriasis
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Does weight decrease the amount of UVB needed to clear psoriasis | 12 weeks
  3 cohorts, all get UVB thrice per week one cohort placebo diet one cohort south beach diet one cohort ornish diet I evaluated PASI 75 improvement within each cohort 0 Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, Principal Investigator — Psoriasis Treatment Center of Central New Jersey